CLINICAL TRIAL: NCT00876135
Title: Role of Airway Hyperresponsiveness on Performance in Elite Swimmers: Efficiency of a Bronchodilator to Prevent an Exercise-induced Bronchoconstriction
Brief Title: Role of Airway Hyperresponsiveness on Performance in Elite Swimmers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Louis-Philippe Boulet, MD, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: proto nage 2
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Inhaled Bronchodilator (Placebo Comparator)
  Interventions: Drug: Ventolin

INTERVENTIONS:
Drug: Ventolin — Ventolin or Placebo will be given before the 4 field tests (2 with ventolin in prevention and 2 with placebo in prevention) and 2 eucapnic voluntary hyperpnoea tests (one preceded by Ventolin and one preceded by Placebo).
  Other Names: Ventolin (salbutamol)

SUMMARY:
The prevalence of airway hyperresponsiveness (AHR) is very high in elite swimmers, reaching 80% in certain studies. Repeated Chlorine-derivatives exposure may be a major causative factor for its development. Asthma diagnosis is generally made on the basis of clinical characteristics. The demonstration of a variable bronchial obstruction through positive expiratory flow reversibility to a bronchodilator, spontaneous variations of airway obstruction or a positive provocation test (methacholine, eucapnic voluntary hyperpnoea…) is necessary to avoid false diagnosis. Currently asthma treatment in swimmers is the same as in the general population. A short-acting bronchodilator is often prescribed to avoid occasional symptoms, combined with an inhaled corticosteroid or an antagonist of Leukotriene if asthma symptoms are persistent. Previous studies have shown a reduced efficiency for asthma medication in elite athletes compared with non-athletes. The specific response to different medications remains to be studied in athletes. The effects of a short-acting bronchodilator in swimmers with AHR, especially when asymptomatic, on pulmonary function and performance have not yet been studied. Moreover, the significance of a positive bronchial provocation test remains to be studied in asymptomatic swimmers with AHR.

DETAILED DESCRIPTION:
Our hypothesis is that swimmers with a positive bronchial provocation challenge have not necessarily an exercise-induced bronchoconstriction during swimming and the use of a bronchodilator will be unnecessary. Chlorine-derivatives exposure may be responsible for a weakness of the epithelium layer but warm and humid atmosphere of the swimming-pools may be protective for the development of a bronchoconstriction. Thus we also hypothesis that during a field test outside the swimming pool, swimmers will develop an exercise-induced asthma, and will need to take a bronchodilator in prevention.

ELIGIBILITY:
Inclusion Criteria:

* Swimmer (at least 10h/week) aged from at least 14 years.

Exclusion Criteria:

* Smoker, obese or other disease which may interfere with the study. Some parts of the study may exclude swimmers taking inhaled corticosteroids.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Bronchodilator versus placebo effects on performance | march to may 2009/ 8 visits

SECONDARY OUTCOMES:
Measurement of oxidative stress | april to June 2009/ 3 visits

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulet, MD, Principal Investigator — Laval University
Locations (1):
- Institut Universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada